CLINICAL TRIAL: NCT00580125
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Fixed Dose, Parallel Group, 3-Week Inpatient Treatment Study To Evaluate The Dose-Response Relationship, Safety, Efficacy, And Pharmacokinetics Of PF-00217830 Compared With Placebo, Using Aripiprazole As A Positive Control, In The Treatment Of Acute Exacerbation Of Schizophrenia
Brief Title: Dose-response Study to Evaluate Safety, Efficacy, and Pharmacokinetics of PF-00217830 Compared With Placebo in Acute Exacerbation of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A7251006
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — PF 00217830; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- A2 (Experimental)
  Interventions: Drug: PF-00217830
- A5 (Placebo Comparator)
  Interventions: Other: Placebo
- A4 (Active Comparator)
  Interventions: Drug: Aripiprazole
- A3 (Experimental)
  Interventions: Drug: PF-00217830
- A1 (Experimental)
  Interventions: Drug: PF-00217830

INTERVENTIONS:
Drug: PF-00217830 — PF-00217830 5 mg, oral capsule, once daily for 21 days
  Arms: A2
Other: Placebo — Placebo, oral capsule, once daily for 21 days
  Arms: A5
Drug: Aripiprazole — Aripiprazole 15 mg, oral capsule, once daily for 21 days
  Other Names: Abilify
  Arms: A4
Drug: PF-00217830 — PF-00217830 15 mg, oral capsule, once daily for 21 days
  Arms: A3
Drug: PF-00217830 — PF-00217830 2 mg, oral capsule, once daily for 21 days
  Arms: A1

SUMMARY:
The objective of this study is demonstrate efficacy and a dose-response in the treatment of acute exacerbation of schizophrenia in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria include:

* Have a current diagnosis of schizophrenia.
* Increase in symptoms over the past 2-4 weeks.
* Willing to remain inpatients for the duration of the trial.

Exclusion Criteria:

* Subjects with a current DSM-IV axis I diagnosis other than schizophrenia
* Subjects who meet the DSM-IV criteria for psychoactive substance abuse and dependence
* Subjects with a history of treatment resistant schizophrenia
* Females of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Clinical laboratory (Screening, Days 1, 7, 14, 21 and Followup); Fasting insulin, HDL, LDL, HbA1c , prolactin, ACTH, and cortisol (Days 1 and 21). | 5 weeks
Physical examination (Screening, Days 1 and 21), neurological examination (Days 1 and 21), and ECG (Screening, Days 1, 7, 14, 20, 21 and Followup). | 5 weeks
Positive and Negative Symptom Scale (PANSS) total score. | Screening, Day 1, 3, 7, 14 and 21
Adverse events (Daily), weight (Screening, Days 1, and 21) and girth (Days 1 and 21), vital signs (Screening, Days 1, 3, 7, 14, 21 and Followup), | 5 weeks
Extrapyramidal Symptom Rating Scale (Screening, Days 1, 3, 7, 14 and 21) and the Stanford Sleepiness Scale (Days 1, 3, 7, 14 and 21). | 4 weeks

SECONDARY OUTCOMES:
PANSS-derived Marder factor scores (positive, negative, disorganized thought, hostility/excitement, anxiety/depression) | Screening, Day 1, 3, 7, 14 and 21
PANSS positive, negative, and general psychopathology subscales | Screening, Day 1, 3, 7, 14 and 21
Clinical Global Impression Scale-S (severity), and Clinical Global Impression Scale-I (improvement) | Screening and Days 1, 3, 7, 14 and 21
NOSIE-30 subscales (irritability, manifest psychosis, personal neatness, retardation, social competence, and social interest) and the GAF. | Days 1 and 21
Treatment Satisfaction Questionnaire for Medication (TSQM) | Day 21
Pharmacokinetics | Days 7, 14, 20, 21, before discharge and Followup
PANSS-derived BPRS core psychosis items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content) | Screening and Days 1, 3, 7, 14 and 21

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (8):
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Bridgeton, Missouri
  - Pfizer Investigational Site, Florissant, Missouri
  - Pfizer Investigational Site, Saint Charles, Missouri
  - Pfizer Investigational Site, Brooklyn, New York
- India (5):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Udupi, Karnataka
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Pune
- Russia (4):
  - Pfizer Investigational Site, Gatchina District, Leningradskaya Oblast'
  - Pfizer Investigational Site, Khot'kovo
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Ukraine (7):
  - Pfizer Investigational Site, Simferopol, Autonomous Republic of Crimea
  - Pfizer Investigational Site, Kiev, Ukraine
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Luhansk

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7251006&StudyName=Dose-response%20study%20to%20evaluate%20safety%2C%20efficacy%2C%20and%20pharmacokinetics%20of%20PF-00217830%20compared%20with%20placebo%20in%20acute%20exacerbation%20of%20sch